CLINICAL TRIAL: NCT05770271
Title: A Novel Electrolyzed Water Spray Reduces the Itching Scores of Patients With Mild Senile Groin Eczema, Neurodermatitis and Psoriasis: A Clinical Study
Brief Title: The Novel Electrolyzed Water Spray Treatment Mild Senile Groin Eczema, Neurodermatitis and Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jia19960129
Record Dates: First submitted 2023-02-26; First posted 2023-03-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Groin Infection; Neurodermatitis; Psoriasis; Eczema
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Itching
MeSH Terms: conditions — Neurodermatitis; Psoriasis; Eczema; Pruritus

STUDY DESIGN:
Masking Description: An open label, single arm and before and after treatment comparison study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The mild senile groin eczema, neurodermatitis and psoriasis and one treatment (Experimental): Participants with itching of mild senile groin eczema, neurodermatitis and psoriasis will receive one treatment with the device and complete the questionnaire.
  Interventions: Device: The novel electrolyzed water spray

INTERVENTIONS:
Device: The novel electrolyzed water spray — Study staff will use the novel electrolyzed water spray device and spray for approximately 5 minutes on the participant's diseased area until half a bottle (200ml) of water is used. The patients use electrolyzed water to treat the diseased area, two times a day, for 10 days. The trial consists of 10 study visits (day 1-day 10). The relief of mild senile groin eczema, neurodermatitis and psoriasis evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.

SUMMARY:
The purpose of this study is to test whether spraying the itching of inflammation skin and groin patients by use of the novel electrolyzed water spray will produce improvement in the condition of itching.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U). This is an open-label, single-arm, and before and after treatment comparison study. This study uses this novel electrolyzed water device and the water spray to treat mild senile groin eczema, neurodermatitis and psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* mild senile groin eczema, neurodermatitis and psoriasis.

Exclusion Criteria:

* severe senile groin eczema, neurodermatitis and psoriasis.
* people with cognitive disorders.
* 80 years or older.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
An itching scale made by modifying the Numeric Pain Rating Scale (NPRS) | 1 hour
  This Score is based on descriptions of the itching that patients rate 0-10 to assess the condition of their itching. A higher score means a worse outcome. 0 means "no itching " and 10 means "the most itching".

SECONDARY OUTCOMES:
A skin signs scale made by modifying the Numeric Pain Rating Scale (NPRS). | 10 days
  The signs of skin chronic inflammation include darkness or redness, swelling and dryness and broken surface and reduced area of the diseased skin. This Score is based on descriptions of signs of senile groin eczema, neurodermatitis and psoriasis rated 0-10 to assess the condition of mild inflammation of the skin and groin. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted